CLINICAL TRIAL: NCT06789224
Title: Validation Study on the Removal of EpCAM-positive Tumour Cells From Blood Collected During Tumour Surgery Using Catumaxomab/Catuvab Device
Acronym: REMOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindis Bloodcare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMOVE
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Bladder Carcinoma; Prostate Tumor; Gallbladder Carcinoma; Endometrial Carcinoma; Gastric Carcinoma; Ovarian Carcinoma; Pancreatic Carcinoma; Colon Carcinoma; Non-small Cell Lung Cancer; Peritoneal Carcinomatosis; Kidney Carcinoma; Liver Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Gallbladder Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Peritoneal Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- medical device validation (Other): removal of tumor cells of EpCAM positive tumors during surgery
  Interventions: Device: CATUVAB

INTERVENTIONS:
Device: CATUVAB — inducing of aggreation of tumor cells and immune cells via trifunctional antibody and removal of aggregates

SUMMARY:
The REMOVE study was an open-label, multicenter validation study on the removal of EpCAM-positive tumor cells from blood collected during tumor surgery using the CATUVAB Kit. The aim of the REMOVE clinical study was to demonstrate the safety and efficacy of the application of the new medical device CATUVAB to allow retransfusion of autologous erythrocyte product produced by an intraoperative blood salvage (IBS) device during oncological high blood loss surgery. The primary objective of the study was to demonstrate that CATUVAB device utilized during autologous blood salvage procedures (including LDFs) depletes intraoperative blood of EpCAM-positive tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Intraoperative blood salvage (IBS)-eligible according to the Investigator
* Patients with a prostate tumor, gallbladder carcinoma, bladder carcinoma, endometrial carcinoma, gastric carcinoma, ovarian carcinoma, pancreatic carcinoma, colon / rectal carcinoma, non-small cell lung cancer, or peritoneal carcinomatosis, i.e., cancer types with a high likelihood of being EpCAM-positive (>92%) OR kidney carcinoma or liver carcinoma.
* For patients with cancer types with a high likelihood of being EpCAM-positive (>92%): if a tumor tissue sample is available and has been EpCAM tested or EpCAM-testing can be done within 5 days of signing the informed consent form (ICF): results of EpCAM typing should be positive.
* For patients with kidney carcinoma or liver carcinoma: a tumor tissue sample must be available and have tested EpCAM-positive prior to surgery.
* Scheduled for surgery to remove tumor.
* The Investigator expects that at least 400 mL full blood can be collected during the tumor surgery.
* An American Society of Anesthesiologists (ASA) Classification of ≤3.

Exclusion Criteria:

* Adjuvant therapy and intra-operative chemotherapy (hyperthermic intraperitoneal hemotherapy, HIPEC) started before blood collection for IBS is completed.
* Lymphocytopenia (count <1.0 x 109 /L lymphocytes).
* Cancer different from indicated types, especially typically EpCAM-negative tumor types.
* Sepsis occurring during surgery.
* Cirrhosis of the liver with a Child-Pugh score of C.
* A thrombocyte count of <30.000/µL.
* Allergies and/or contraindications against Catumaxomab or any of the components or ingredients used in the IBS procedure (e.g., leukocyte depletion filter [LDF], diluent, buffer solution or anticoagulants).
* Active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, confirmed by a positive polymerase chain reaction (PCR) test prior surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
depletion of EpCAM-positive tumor cells | during surgery only
  Tumor cell count (Depletion) measured with Immun-histo chemistry staining and tumor cell counting in a Neubauer Chamber
  * a depletion to ≤10 cells per 100 mL EC, OR
  * if <100.000 tumor cells have been detected before in IBS: a depletion by at least a factor of 103 in the EC (total) as compared to collected intraoperative blood (total), OR
  * if ≥100.000 tumor cells have been detected before in IBS: a depletion by at least a factor of 5x103 in the EC (total) as compared to collected intraoperative blood (total), in at least 95% of subjects after one IBS/LDF cycle using the Catuvab device. The primary endpoint will only be determined in subjects with EpCAM-positive tumor cells in salvaged blood and who receive retransfusion of the EC

CONTACTS AND LOCATIONS:
Overall Officials: Markus Heiss, MD, Study Chair — University Köln Merheim
Locations (6):
- Germany (6):
  - Kliniken der Stadt Köln gGmbH, Cologne, North Rhine-Westphalia
  - Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz Klinik für Anästhesiologie, Mainz
  - Universitätsmedizin Mannheim, Klinik für Urologie und Urochirurgie, Mannheim
  - Klinikum Traunstein, Traunstein
  - Klinik und Poliklinik für Anästhesiologie, Intensivmedizin, Notfallmedizin und Schmerztherapie Universitätsklinikum Würzburg, Würzburg